CLINICAL TRIAL: NCT03480945
Title: Evaluation of the Mechanism Underlying Endothelial Dysfunction in Patients With Type 2 Diabetes With Poor and Optimized Glycaemic Control
Brief Title: Glycemic Control and Endothelial Function in Patients With Type 2 Diabetes
Acronym: AIDdiabetes
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, professor, Karolinska Institutet
Other Study IDs: AIDdiabetes
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serotonin — Endothelium-dependent dilatation
  Other Names: nitroprusside

SUMMARY:
Study objective To evaluate the mechanism behind endothelial dysfunction in patients with type 2 diabetes in relation to the level of glycaemic control.

Primary endpoint: Change in endothelium dependent vasodilatation (EDV).

DETAILED DESCRIPTION:
The study is performed on one group of patients with type 2 diabetes and one group of age-matched healthy controls

Inclusion criteria:

1. Type 2 diabetes
2. Poor glycaemic control defined as a mean day blood glucose >12 mmol/L.

Exclusion criteria:

1. Age >80 years.
2. HbA1c <70 mmol/mol
3. Myocardial infarction/unstable angina within 6 weeks prior to the study.
4. Treatment with oral anticoagulants (Warfarin or New oral anticoagulants)
5. Raynaud's phenomenon, peripheral vasculopathies, arterial shunting or other vascular surgery of the study arm.
6. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.
7. Participant in an ongoing study.
8. Unwillingness to participate following oral and written information.

Healthy controls Inclusion criteria

1. No medical history of cardiovascular disease 2. Fasting blood glucose <6.0 mmol/l or plasma glucose <7.0 mmol/l Exclusion criteria

1. Age >80 years.
2. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.
3. Participant in an ongoing study.
4. Unwillingness to participate following oral and written information.

Endothelium-dependent vasodilatation is determined by venous occlusion plethysmography during intra-arterial infusion of serotonin (21, 70 and 210 ng/min). Endothelium-independent vasodilatation is determined by infusion of sodium nitroprusside (SNP; 1, 3 and 10 µg/min). Each dose is given for 2 min at a rate of 2.5 ml/min.

Sixteen patients and age-matched healthy controls are included. On the day of the study the subject arrives to the laboratory after having a light breakfast. Forearm vessels of the non-dominant arm are cannulated and forearm blood flow is determined as described above. Baseline endothelium dependent and endothelium independent vasodilatation is determined by intra-arterial infusions of serotonin and SNP, respectively, during an intra-arterial infusion of saline. Thereafter an intra-arterial infusion of the arginase inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA) is started and is maintained for 120 min at a rate of 0.1 mg/min. The dose is based on a previous study by our group demonstrating improved endothelial function. Endothelium-dependent and -independent vasodilatation is reassessed at 120 min of infusion.

Following determination of baseline endothelial function (poor glycemic control), the patients are put on optimized glucose lowering therapy with insulin and/or oral glucose lowering medication according to clinical routine at the day-care center of the department of Endocrinology, Karolinska University Hospital for at least 8 weeks. Treatment target is mean day blood glucose <9 mmol/L and fasting blood glucose 4-6 mmol/L. After this, endothelium-dependent and -independent vasodilatation before and following arginase inhibition is re-assessed as described above.The healthy control group is only investigated on one occasion.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Poor glycaemic control defined as a mean day blood glucose >12 mmol/L.

Exclusion Criteria:

1. Age >80 years.
2. HbA1c <70 mmol/mol
3. Myocardial infarction/unstable angina within 6 weeks prior to the study.
4. Treatment with oral anticoagulants (Warfarin or New oral anticoagulants)
5. Raynaud's phenomenon, peripheral vasculopathies, arterial shunting or other vascular surgery of the study arm.
6. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.
7. Participant in an ongoing study.
8. Unwillingness to participate following oral and written information.

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes Healthy controls
Enrollment: 16 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 8 weeks
  Change in endothelium-dependent dilatation

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided